CLINICAL TRIAL: NCT04529746
Title: A Pilot Evaluation of the EVERYbody Project: Professionally-delivered Inclusive Eating Disorder Risk Factor Reduction for College Students
Brief Title: Pilot Evaluation of the EVERYbody Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Washington University (Other)
Responsible Party: Principal Investigator, Anna Ciao, Associate Professor of Psychology, Western Washington University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-004_1
Record Dates: First submitted 2020-08-15; First posted 2020-08-28 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Body Image; Eating Disorder Symptom

STUDY DESIGN:
Intervention Model Description: Participants were randomized on a 1-1 basis to receive either the EVERYbody Project or be on the waitlist control list (assessment-only control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVERYbody Project: Professional facilitator version (Experimental): The EVERYbody Project is a dissonance body image intervention created from focus group feedback (Ciao, Ohls, & Pringle, 2017) and through an iterative process of student-driven feedback. The Body Project manual (Stice et al., 2006) was adapted to retain key dissonance activities while expanding the gender focus, adding an exploration of the diversity characteristics within appearance ideals, and adjusting activities to be inclusive of diversity characteristics. Several adapted versions of the intervention were piloted with groups of college students and further adapted based on feedback.
  Facilitators received 16 hours of training on the EVERYbody Project manual and facilitation guidelines.
  Interventions: Behavioral: EVERYbody Project
- Waitlist control group (No Intervention): Participants allocated to the waitlist completed assessments at time points parallel to those in the EVERYbody Project condition and were offered the EVERYbody Project upon completing the one-month follow-up assessment.

INTERVENTIONS:
Behavioral: EVERYbody Project — Brief behavioral intervention (4 hours across two meetings)
  Arms: EVERYbody Project: Professional facilitator version

SUMMARY:
A pilot randomized-controlled trial explored the feasibility, acceptability, and efficacy of an inclusive dissonance-based body image intervention called the EVERYbody Project. The professionally delivered EVERYbody Project was evaluated in a universal college student population compared to a waitlist control group through one-month follow-up.

DETAILED DESCRIPTION:
An existing dissonance-based body image program (the Body Project; Stice, Shaw, Burton, & Wade, 2006) was adapted to directly discuss diversity within cultural appearance ideals (including race, gender identity, sexuality, ability, and age) and the individual and collective impact of pursuing exclusive appearance norms.

The feasibility, acceptability, and efficacy of the EVERYbody Project was assessed in an initial randomized-controlled trial. College students within a university in the Pacific Northwest United States were invited to participate in programming (universal intervention target).

Professional delivery of the two-session EVERYbody Project was compared to a waitlist control condition. Intervention groups were facilitated by one "expert" (faculty or staff with body image expertise) and two college student co-facilitators. Mixed methods assessment included a comparison of changes in quantitative eating disorder risk factor outcomes across randomization conditions and among students with marginalized identities at pre-intervention, post-intervention, and one-month follow-up. Qualitative interviews assessed the impact of the program on participants with marginalized identities. Feasibility and acceptability of the program was assessed to evaluate the appropriateness of the EVERYbody Project within universal college student audiences.

ELIGIBILITY:
Inclusion Criteria:

* Current college student enrolled at institution where research was taking place

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms | Assessed change from baseline (Survey 1) through post-intervention (Survey 2; immediately after intervention) and one-month follow-up (Survey 3; one month after intervention). Waitlist was assessed at parallel time points.
  Eating disorder symptoms were assessed with the Eating Disorders Examination Questionnaire (EDEQ; Fairburn & Beglin, 1994). The Global score of the EDEQ was used in this study (average across all 28 items with a 0-6 range; higher scores equal greater eating disorder symptoms).
Body dissatisfaction: The Satisfaction and Dissatisfaction with Body Parts Scale | Assessed change from baseline (Survey 1) through post-intervention (Survey 2; immediately after intervention) and one-month follow-up (Survey 3; one month after intervention). Waitlist was assessed at parallel time points.
  The Satisfaction and Dissatisfaction with Body Parts Scale (SDBPS; Berscheid, Walster, & Bohrnstedt, 1973) assessed satisfaction and dissatisfaction with nine parts of the body that are commonly endorsed as concerning (e.g., stomach, thighs, hips). The average score was used in this study (average across all 9 items with 1-5 range; higher scores equal greater body dissatisfaction).
Internalized cultural appearance norms | Assessed change from baseline (Survey 1) through post-intervention (Survey 2; immediately after intervention) and one-month follow-up (Survey 3; one month after intervention). Waitlist was assessed at parallel time points.
  The two Internalization subscales of the Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4; Schaefer et al., 2015) assess internalized cultural messages surrounding appearance and attractiveness. The two internalization subscales were combined for this study (average across all 10 items with 1-5 range; higher scores equal greater internalization), following prior research by Kilpela et al. (2016).

SECONDARY OUTCOMES:
Negative affect | Assessed change from baseline (Survey 1) through post-intervention (Survey 2; immediately after intervention) and one-month follow-up (Survey 3; one month after intervention). Waitlist was assessed at parallel time points.
  Negative affect was assessed with 20 items from the fear, guilt, and sadness subscales of the Positive and Negative Affect Schedule-Revised (PANAS-X; Watson & Clark, 1992). The average of all 20 items was used in this study with 1-5 range; higher scores equal greater negative affect.

OTHER OUTCOMES:
Open-ended interviews | Students are invited to participate after completing their follow-up survey (Survey 3) or one month after their participation in the EVERYbody Project.
  Students with marginalized identities who participated in EVERYbody Project groups were invited to complete semi-structured interviews. Specific question asked were:
  1. How was your experience with the EVERYbody Project?
  2. Was anything in the program (any activity or part of the experience) particularly interesting or helpful to you? Why?
  3. Was anything in the program (any activity or part of the experience) particularly unhelpful or upsetting to you? Why?
  (3) The goal of this research was to have conversations about body image that are more inclusive, that is, with diverse individuals who have many different experiences. Do you think this occurred within your EVERYbody Project group? (4) Is there anything you would suggest for improving EVERYbody Project groups to meet the goal stated above? (5) Is there anything else you would like to share with us about the EVERYbody Project?
  Additional follow-up prompts were used at the interviewer's discretion.
Program satisfaction and application: questions included four Likert scale | Assessed at post-intervention (Survey 2; immediately following the intervention) and one-month follow-up (Survey 3; four weeks post intervention).
  Satisfaction with the EVERYbody Project (based on Ciao et al., 2015) included four Likert scale items (e.g., "I enjoyed the EVERYbody Project") rated from 1 (strongly disagree) to 5 (strongly agree). Questions were averaged to create a total "satisfaction" score; higher scores equaled greater satisfaction. Open-ended questions also assessed satisfaction (e.g., "Was any part of the EVERYbody Project particularly helpful/useful? If so, which part and why?"). Satisfaction questions were administered immediately following participation in the intervention (Survey 2).
  At post-intervention (Survey 2) and one-month follow-up (Survey 3), three questions gauged application of information learned in the program (e.g., "How often do think about the things you learned in the EVERYbody Project?" rated on a scale from 1 (not at all) to 5 (all the time). Items were averaged to created a total "application" score with higher scores equaling greater application of intervention content.

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Ciao, PhD, Principal Investigator — Western Washington University
Locations (1):
- Western Washington University, Bellingham, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and other materials will be made available following reasonable request to study Principal Investigator. All outcome data will be included in data sharing. Socio-demographic characteristics will be collapsed into broader categories to protect participant identity.
  Other study materials, including intervention manuals, will be housed on the Principal Investigator's Open Science Framework page, where URLs will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the trial is complete, data are available immediately upon request.
URL: https://osf.io/x3k7v/?view_only=c9dbd31a4ad94a08b16421d719bc0fac

REFERENCES:
- [Background] Ciao AC, Ohls OC, Pringle KD. Should body image programs be inclusive? A focus group study of college students. Int J Eat Disord. 2018 Jan;51(1):82-86. doi: 10.1002/eat.22794. Epub 2017 Nov 6. PMID 29105805
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Background] Berscheid, E., Hatfield [Walster], E., & Bohrnstedt, G. (1973). The happy American body: A survey report. Psychology Today, 7, 119-131.
- [Background] Watson, D., & Clark, L. A. (1992). Affects separable and inseparable: On the hierarchical arrangement of the negative affects. Journal of Personality and Social Psychology, 62, 489-505. http://dx.doi.org/10.1037/ 0022-3514.62.3.489
- [Background] Ciao AC, Latner JD, Brown KE, Ebneter DS, Becker CB. Effectiveness of a peer-delivered dissonance-based program in reducing eating disorder risk factors in high school girls. Int J Eat Disord. 2015 Sep;48(6):779-84. doi: 10.1002/eat.22418. Epub 2015 May 8. PMID 25959408
- [Background] Kilpela LS, Blomquist K, Verzijl C, Wilfred S, Beyl R, Becker CB. The body project 4 all: A pilot randomized controlled trial of a mixed-gender dissonance-based body image program. Int J Eat Disord. 2016 Jun;49(6):591-602. doi: 10.1002/eat.22562. Epub 2016 May 18. PMID 27188688
- [Result] Ciao AC, Munson BR, Pringle KD, Roberts SR, Lalgee IA, Lawley KA, Brewster J. Inclusive dissonance-based body image interventions for college students: Two randomized-controlled trials of the EVERYbody Project. J Consult Clin Psychol. 2021 Apr;89(4):301-315. doi: 10.1037/ccp0000636. PMID 34014692